CLINICAL TRIAL: NCT03667404
Title: Gut Microbial Remodeling with Resistant Maltodextrin for Motor and Non-motor Symptoms in Parkinson's Disease: Safety and Tolerability Study
Brief Title: Resistant Maltodextrin for Gut Microbiome in Parkinson's Disease: Safety and Tolerability Study
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Roneil Malkani, Assistant Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STU00207142
Record Dates: First submitted 2018-09-10; First posted 2018-09-12 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2024-02

CONDITIONS: Parkinson Disease; Intestinal Bacteria Flora Disturbance; Dietary Modification
Keywords: Resistant maltodextrin; dietary fiber; gut microbiome; Parkinson's disease
MeSH Terms: conditions — Parkinson Disease | interventions — maltodextrin

STUDY DESIGN:
Intervention Model Description: Double blind placebo (maltodextrin) controlled randomized trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: participants will be blinded to condition. control condition (maltodextrin) will be used and has identical appearance.
  investigator and research staff (except pharmacy) will be blinded to condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Resistant Maltodextrin (Experimental): Resistant maltodextrin (RM) powder 25 g during days 1-7 and 50g during days 8-28, each dose dissolved in 8 oz of water once daily in the morning.
  Interventions: Dietary Supplement: Resistant maltodextrin
- Maltodextrin (Placebo Comparator): Maltodextrin 25g for days 1-7 and 50 g for days 8-28, each dose dissolved in 8 oz of water once daily in the morning.
  Interventions: Dietary Supplement: maltodextrin

INTERVENTIONS:
Dietary Supplement: Resistant maltodextrin — Resistant maltodextrin powder
  Arms: Resistant Maltodextrin
Dietary Supplement: maltodextrin — maltodextrin powder
  Arms: Maltodextrin

SUMMARY:
This study will evaluate the safety and tolerability of a dietary fiber, resistant maltodextrin, in people with Parkinson's disease. It will also evaluate the fiber's effect on the gut microbiome and potential effects on motor function and non-motor functions. Half of the participants will receive resistant maltodextrin and the other half will receive a control substance, maltodextrin.

DETAILED DESCRIPTION:
Intestinal microbiota may play in important role in Parkinson's disease (PD). Colonic bacteria play roles in multiple functions including gut motility and secretion of metabolites which can have systemic effects on the body. Recent evidence has shown that people with PD have an altered distribution of gut bacteria that healthy controls. These changes are associated with differences in various metabolites, including butyrate, that are involved in maintaining the gut barrier integrity and even gait and balance function. Microbiota dysbiosis could potentially exacerbate or even contribute to the pathogenesis of PD. Probiotic and dietary interventions may improve gut function and the motor symptoms in PD, but neither have been examined for their effect on the gut microbiome. Prebiotic treatments have been shown to order the microbiome in some populations, but have not been assessed for tolerability or efficacy in PD.

The objective of this study is to examine the safety and tolerability of resistant maltodextrin (RM), a prebiotic non-digestible fiber, and its effect on the microbiome and motor in non-motor symptoms and PD. The investigators will conduct a randomized, parallel-group double-blinded controlled trial assessing RM 50 g daily compared to maltodextrin (an easily digestible glucose polysaccharide) over 4 weeks. Patients will be dosed with 25 g daily for 1 week and then titrated to 50 g daily for the remaining 3 weeks.

The goals of this study include: 1) To determine the safety and tolerability of RM compared to maltodextrin in patients with PD; 2) To determine if RM will remodel the gut microbiome in patients with PD; 3) (exploratory) To determine if RM administration will improve motor and non-motor symptoms in PD.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age ≥60 years
* Diagnosis of PD based on United Kingdom PD brain bank criteria, Hoehn and Yahr stage 1-3.
* Stable dose of PD medications for 30 days prior to study and for duration of study
* If used, stable dose of melatonin, sedative/hypnotic or stimulant medications

Exclusion Criteria:

* use of other prebiotic or probiotic treatment for 30 days prior to or during the study
* unstable medical or psychiatric disorder
* history of diabetes mellitus or current use of medication for diabetes
* cognitive impairment based on Montreal Cognitive Assessment (MoCA) <25.
* current or recent (within previous 3 weeks) use of laxatives
* use of antibiotics in the past 30 days
* participation in another clinical trial in the past 30 days.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-11-06 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 4 weeks
  Adverse event frequency and severity based on diary reports, phone calls, and in-person assessments.

SECONDARY OUTCOMES:
Gut microbial remodeling | 4 weeks
  Change in fecal butyrate-producing bacteria based on high-throughput amplicon sequencing of the V4 variable region of the microbial 16s ribosomal ribonucleic acid (RNA) gene.

CONTACTS AND LOCATIONS:
Overall Officials: Roneil G Malkani, Principal Investigator — Northwestern Feinberg School of Medicine Department of Neurology
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baer DJ, Stote KS, Henderson T, Paul DR, Okuma K, Tagami H, Kanahori S, Gordon DT, Rumpler WV, Ukhanova M, Culpepper T, Wang X, Mai V. The metabolizable energy of dietary resistant maltodextrin is variable and alters fecal microbiota composition in adult men. J Nutr. 2014 Jul;144(7):1023-9. doi: 10.3945/jn.113.185298. Epub 2014 Apr 17. PMID 24744316
- [Background] Braak H, Rub U, Gai WP, Del Tredici K. Idiopathic Parkinson's disease: possible routes by which vulnerable neuronal types may be subject to neuroinvasion by an unknown pathogen. J Neural Transm (Vienna). 2003 May;110(5):517-36. doi: 10.1007/s00702-002-0808-2. PMID 12721813
- [Background] Cassani E, Privitera G, Pezzoli G, Pusani C, Madio C, Iorio L, Barichella M. Use of probiotics for the treatment of constipation in Parkinson's disease patients. Minerva Gastroenterol Dietol. 2011 Jun;57(2):117-21. PMID 21587143
- [Background] Fastinger ND, Karr-Lilienthal LK, Spears JK, Swanson KS, Zinn KE, Nava GM, Ohkuma K, Kanahori S, Gordon DT, Fahey GC Jr. A novel resistant maltodextrin alters gastrointestinal tolerance factors, fecal characteristics, and fecal microbiota in healthy adult humans. J Am Coll Nutr. 2008 Apr;27(2):356-66. doi: 10.1080/07315724.2008.10719712. PMID 18689571
- [Background] Forsyth CB, Shannon KM, Kordower JH, Voigt RM, Shaikh M, Jaglin JA, Estes JD, Dodiya HB, Keshavarzian A. Increased intestinal permeability correlates with sigmoid mucosa alpha-synuclein staining and endotoxin exposure markers in early Parkinson's disease. PLoS One. 2011;6(12):e28032. doi: 10.1371/journal.pone.0028032. Epub 2011 Dec 1. PMID 22145021
- [Background] Hawkes CH, Del Tredici K, Braak H. Parkinson's disease: a dual-hit hypothesis. Neuropathol Appl Neurobiol. 2007 Dec;33(6):599-614. doi: 10.1111/j.1365-2990.2007.00874.x. Epub 2007 Oct 24. PMID 17961138
- [Background] He B, Nohara K, Ajami NJ, Michalek RD, Tian X, Wong M, Losee-Olson SH, Petrosino JF, Yoo SH, Shimomura K, Chen Z. Transmissible microbial and metabolomic remodeling by soluble dietary fiber improves metabolic homeostasis. Sci Rep. 2015 Jun 4;5:10604. doi: 10.1038/srep10604. PMID 26040234
- [Background] Holmqvist S, Chutna O, Bousset L, Aldrin-Kirk P, Li W, Bjorklund T, Wang ZY, Roybon L, Melki R, Li JY. Direct evidence of Parkinson pathology spread from the gastrointestinal tract to the brain in rats. Acta Neuropathol. 2014 Dec;128(6):805-20. doi: 10.1007/s00401-014-1343-6. Epub 2014 Oct 9. PMID 25296989
- [Background] Keshavarzian A, Green SJ, Engen PA, Voigt RM, Naqib A, Forsyth CB, Mutlu E, Shannon KM. Colonic bacterial composition in Parkinson's disease. Mov Disord. 2015 Sep;30(10):1351-60. doi: 10.1002/mds.26307. Epub 2015 Jul 16. PMID 26179554
- [Background] Kishimoto Y, Kanahori S, Sakano K, Ebihara S. The maximum single dose of resistant maltodextrin that does not cause diarrhea in humans. J Nutr Sci Vitaminol (Tokyo). 2013;59(4):352-7. doi: 10.3177/jnsv.59.352. PMID 24064737
- [Background] Lee A, Gilbert RM. Epidemiology of Parkinson Disease. Neurol Clin. 2016 Nov;34(4):955-965. doi: 10.1016/j.ncl.2016.06.012. Epub 2016 Aug 18. PMID 27720003
- [Background] Li S, Wang Y, Wang F, Hu LF, Liu CF. A New Perspective for Parkinson's Disease: Circadian Rhythm. Neurosci Bull. 2017 Feb;33(1):62-72. doi: 10.1007/s12264-016-0089-7. Epub 2016 Dec 19. PMID 27995565
- [Background] Martinez-Martin P. The importance of non-motor disturbances to quality of life in Parkinson's disease. J Neurol Sci. 2011 Nov 15;310(1-2):12-6. doi: 10.1016/j.jns.2011.05.006. Epub 2011 May 31. PMID 21621226
- [Background] Miyazato S, Kishimoto Y, Takahashi K, Kaminogawa S, Hosono A. Continuous intake of resistant maltodextrin enhanced intestinal immune response through changes in the intestinal environment in mice. Biosci Microbiota Food Health. 2016;35(1):1-7. doi: 10.12938/bmfh.2015-009. Epub 2015 Aug 25. PMID 26858925
- [Background] Nagahara AH, Tuszynski MH. Potential therapeutic uses of BDNF in neurological and psychiatric disorders. Nat Rev Drug Discov. 2011 Mar;10(3):209-19. doi: 10.1038/nrd3366. PMID 21358740
- [Background] Pan-Montojo F, Schwarz M, Winkler C, Arnhold M, O'Sullivan GA, Pal A, Said J, Marsico G, Verbavatz JM, Rodrigo-Angulo M, Gille G, Funk RH, Reichmann H. Environmental toxins trigger PD-like progression via increased alpha-synuclein release from enteric neurons in mice. Sci Rep. 2012;2:898. doi: 10.1038/srep00898. Epub 2012 Nov 30. PMID 23205266
- [Background] Perez-Pardo P, de Jong EM, Broersen LM, van Wijk N, Attali A, Garssen J, Kraneveld AD. Promising Effects of Neurorestorative Diets on Motor, Cognitive, and Gastrointestinal Dysfunction after Symptom Development in a Mouse Model of Parkinson's Disease. Front Aging Neurosci. 2017 Mar 20;9:57. doi: 10.3389/fnagi.2017.00057. eCollection 2017. PMID 28373840
- [Background] Queipo-Ortuno MI, Seoane LM, Murri M, Pardo M, Gomez-Zumaquero JM, Cardona F, Casanueva F, Tinahones FJ. Gut microbiota composition in male rat models under different nutritional status and physical activity and its association with serum leptin and ghrelin levels. PLoS One. 2013 May 28;8(5):e65465. doi: 10.1371/journal.pone.0065465. Print 2013. PMID 23724144
- [Background] Sampson TR, Debelius JW, Thron T, Janssen S, Shastri GG, Ilhan ZE, Challis C, Schretter CE, Rocha S, Gradinaru V, Chesselet MF, Keshavarzian A, Shannon KM, Krajmalnik-Brown R, Wittung-Stafshede P, Knight R, Mazmanian SK. Gut Microbiota Regulate Motor Deficits and Neuroinflammation in a Model of Parkinson's Disease. Cell. 2016 Dec 1;167(6):1469-1480.e12. doi: 10.1016/j.cell.2016.11.018. PMID 27912057
- [Background] Savignac HM, Corona G, Mills H, Chen L, Spencer JP, Tzortzis G, Burnet PW. Prebiotic feeding elevates central brain derived neurotrophic factor, N-methyl-D-aspartate receptor subunits and D-serine. Neurochem Int. 2013 Dec;63(8):756-64. doi: 10.1016/j.neuint.2013.10.006. Epub 2013 Oct 16. PMID 24140431
- [Background] Scheperjans F, Aho V, Pereira PA, Koskinen K, Paulin L, Pekkonen E, Haapaniemi E, Kaakkola S, Eerola-Rautio J, Pohja M, Kinnunen E, Murros K, Auvinen P. Gut microbiota are related to Parkinson's disease and clinical phenotype. Mov Disord. 2015 Mar;30(3):350-8. doi: 10.1002/mds.26069. Epub 2014 Dec 5. PMID 25476529
- [Background] Tandberg E, Larsen JP, Karlsen K. A community-based study of sleep disorders in patients with Parkinson's disease. Mov Disord. 1998 Nov;13(6):895-9. doi: 10.1002/mds.870130606. PMID 9827612
- [Background] Thaiss CA, Zeevi D, Levy M, Zilberman-Schapira G, Suez J, Tengeler AC, Abramson L, Katz MN, Korem T, Zmora N, Kuperman Y, Biton I, Gilad S, Harmelin A, Shapiro H, Halpern Z, Segal E, Elinav E. Transkingdom control of microbiota diurnal oscillations promotes metabolic homeostasis. Cell. 2014 Oct 23;159(3):514-29. doi: 10.1016/j.cell.2014.09.048. Epub 2014 Oct 16. PMID 25417104
- [Background] Tomlinson CL, Stowe R, Patel S, Rick C, Gray R, Clarke CE. Systematic review of levodopa dose equivalency reporting in Parkinson's disease. Mov Disord. 2010 Nov 15;25(15):2649-53. doi: 10.1002/mds.23429. PMID 21069833
- [Background] Unger MM, Moller JC, Mankel K, Eggert KM, Bohne K, Bodden M, Stiasny-Kolster K, Kann PH, Mayer G, Tebbe JJ, Oertel WH. Postprandial ghrelin response is reduced in patients with Parkinson's disease and idiopathic REM sleep behaviour disorder: a peripheral biomarker for early Parkinson's disease? J Neurol. 2011 Jun;258(6):982-90. doi: 10.1007/s00415-010-5864-1. Epub 2010 Dec 24. PMID 21181542
- [Background] Unger MM, Spiegel J, Dillmann KU, Grundmann D, Philippeit H, Burmann J, Fassbender K, Schwiertz A, Schafer KH. Short chain fatty acids and gut microbiota differ between patients with Parkinson's disease and age-matched controls. Parkinsonism Relat Disord. 2016 Nov;32:66-72. doi: 10.1016/j.parkreldis.2016.08.019. Epub 2016 Aug 26. PMID 27591074
- [Background] Wallace CJK, Milev R. The effects of probiotics on depressive symptoms in humans: a systematic review. Ann Gen Psychiatry. 2017 Feb 20;16:14. doi: 10.1186/s12991-017-0138-2. eCollection 2017. PMID 28239408